CLINICAL TRIAL: NCT04100031
Title: Efficacy of an Ocular Bandage Contact Lens for the Treatment of Dry Eye After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuwen2018-082
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-01

CONDITIONS: Cataract; Dry Eye
MeSH Terms: conditions — Cataract; Dry Eye Syndromes | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCL group (Experimental)
  Interventions: Device: bandage contact lenses; Procedure: phacoemulsification
- control group (Active Comparator)
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Device: bandage contact lenses — wear bandage contact lensesfor a week after cataract surgery.
  Arms: BCL group
Procedure: phacoemulsification — underwent standard phacoemulsification through a 2.8-mm clear corneal temporal incision and intraocular lens

SUMMARY:
To study the efficacy of an ocular bandage contact lens for the treatment of dry eye after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

1. age-related cataract
2. dry eye disease

Exclusion Criteria:

1. a history of surgery and other ocular diseases
2. contact lens use
3. ocular therapies such as 0.05% cyclosporine A or steroids in the last 3 months. had 4.any systemic diseases such as heart diseases, diabetes and psychosis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Ocular Surface Disease Index at 1 week | 0 day, 1 week postoperative
  Ocular Surface Disease Index
Change from Baseline Ocular Surface Disease Index at 1 month | 0 day, 1 month postoperative
  Ocular Surface Disease Index
Change from Baseline meibography score at 1 week | 0 day, 1 week postoperative
  meibography score
Change from Baseline meibography score at 1 month | 0 day, 1 month postoperative
  meibography score
Change from Baseline of non-invasive keratograph tear meniscus height at 1 month | 0 day, 1 month postoperative
  non-invasive keratograph tear meniscus height
Change from Baseline of non-invasive keratograph tear meniscus height at 1 week | 0 day, 1 week postoperative
  non-invasive keratograph tear meniscus height
Change from Baseline noninvasive tear breakup time at 1 week | 0 day, 1 week postoperative
  noninvasive tear breakup time
Change from Baseline noninvasive tear breakup time at 1 month | 0 day, 1 month postoperative
  noninvasive tear breakup time
Change from Baseline Schirmer I test at 1 week | 0 day, 1 week postoperative
  Schirmer I test
Change from Baseline Schirmer I test at 1 month | 0 day, 1 month postoperative
  Schirmer I test
slit-lamp examination | 0 day
  slit-lamp examination
Change from Baseline IL-1, IL-6, IL-12, IL-10, IL-8, TNF-α and ICAM-1 level at 1 month | 0 day and 1 month postoperative
  cytokine levels

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wu X, Ma Y, Chen X, He S, Lin X, Yu X, Chen W, Luo C, Xu W. Efficacy of bandage contact lens for the management of dry eye disease after cataract surgery. Int Ophthalmol. 2021 Apr;41(4):1403-1413. doi: 10.1007/s10792-021-01692-6. Epub 2021 Jan 28. PMID 33507461